CLINICAL TRIAL: NCT03933878
Title: Rapid Detection of Airway Pathogens for Lung Transplantation
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: BioFire Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P0535801
Record Dates: First submitted 2019-04-24; First posted 2019-05-01 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Lung Transplantation; Respiratory Tract Infections; Pulmonary Infection
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Post-transplant recipient BAL samples: No intervention will be administered
- Donor BAL samples: No intervention will be administered

SUMMARY:
Pneumonias and lower respiratory tract infections can have important long-term consequences, particularly in the context of lung transplantation, where pneumonia is a major cause of death. Candidate organs and lung transplant recipients undergo bronchoscopic inspection to assess for lower respiratory tract infection, but traditional culture methods take time, leading to increased risk from inappropriate therapy. The investigators hypothesize that the rapid detection of lower respiratory tract infection, using a semi-quantitative multiplex molecular assay, can decrease the time to appropriate clinical decision making.

DETAILED DESCRIPTION:
Before and after lung transplantation, clinical decision-making for infection diagnosis can be delayed by the time requirements of traditional culture techniques. This study will enroll lung transplant donor candidates and recipients undergoing assessment for lower respiratory tract infection by bronchoscopic alveolar lavage (or washing). The investigators will record bronchoscopy time and time to test result and clinical management decision based on traditional culture methods. The investigators will perform a semi-quantitative multiplex molecular assay for lower respiratory tract infection using the BioFire Pneumonia Panel and these results will be evaluated by clinicians not directly involved in patient care. Timing and outcome of clinical decision making will be recorded. The investigators will compare the time to result using a paired Student's t-test between traditional and molecular methods. Secondary endpoints include time to clinical decision, postulated changes in clinical decisions, and agreement between methods.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be included if subjects are able and willing to provide informed consent for this study as part of an ongoing prospective biorepository and clinical data repository cohort study.
* Donors can be included as subjects if families provide informed consent.

Exclusion Criteria:

* Samples from donor organs will be excluded if the organs are unlikely likely to be used based on review of preliminary data.
* Post-transplant samples will be excluded if the suspicion for infection is sufficiently low that lavage samples are not sent for microbiologic workup or there is insufficient sample for research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve adult lung transplant donors and recipients at UCSF.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Time to result | One year
  The investigators will measure the difference between the time that microbiology results became available using standard of care diagnostics and the time of result from molecular methods.

SECONDARY OUTCOMES:
Changes in clinical management or treatment | One year
  The investigators will record clinical management decisions resulting from both the BioFire molecular diagnostic assay and the current standard of care clinical procedures. The study will report the percentage agreement on treatment decisions between the two diagnostic pathways.
Agreement between assays | One year
  The investigators will record pathogen detection results from both the BioFire molecular diagnostic assay and the current standard of care clinical procedures. The investigators will then report the percentage agreement on pathogen detection between the two diagnostic pathways.

CONTACTS AND LOCATIONS:
Overall Officials: John Greenland, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Parnassus, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No